CLINICAL TRIAL: NCT02555540
Title: Clinical Study to Generate a Set of Data Characterising Clinical Events, Physiological Responses, and Innate and Adaptive Immune Responses Following a Single IM Immunisation With Boostrix® or Placebo in Healthy Adults
Brief Title: Placebo Controlled Study to Generate Data Characterising Safety Parameters and Immune Responses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University of Surrey (Other); Novartis Vaccines (Industry); Max Planck Institute for Infection Biology (Other); deCODE genetics (Industry); GlaxoSmithKline (Industry); Sanofi Pasteur, a Sanofi Company (Industry); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BioVacSafe - Boostrix
Record Dates: First submitted 2015-08-24; First posted 2015-09-21 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Prevention of Infections With Bordetella Pertussis
MeSH Terms: interventions — Boostrix; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (16):
- Boostrix, Male, >/= 5 years, D2 visit (Active Comparator): 25 male subjects who have received their last dT(Pa) vaccine at least 5 years ago, and who have the Visit 2 on 'Day 2'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 2 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Boostrix
- Boostrix, Male, >/= 5 years, D3 visit (Active Comparator): 25 male subjects who have received their last dT(Pa) vaccine at least 5 years ago, and who have the Visit 2 on 'Day 3'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Boostrix
- Boostrix, Female, >/= 5 years, D2 visit (Active Comparator): 25 female subjects who have received their last dT(Pa) vaccine at least 5 years ago, and who have the Visit 2 on 'Day 2'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 2 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Boostrix
- Boostrix, Female, >/= 5 years, D3 visit (Active Comparator): 25 female subjects who have received their last dT(Pa) vaccine at least 5 years ago, and who have the Visit 2 on 'Day 3'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Boostrix
- Placebo, Male, >/= 5 years, D2 visit (Placebo Comparator): 5 male subjects who have received their last dT(Pa) vaccine at least 5 years ago, and who have the Visit 2 on 'Day 2'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 2 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Placebo (Saline)
- Placebo, Male, >/= 5 years, D3 visit (Placebo Comparator): 5 male subjects who have received their last dT(Pa) vaccine at least 5 years ago, and who have the Visit 2 on 'Day 3'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Placebo (Saline)
- Placebo, Female, >/= 5 years, D2 visit (Placebo Comparator): 5 female subjects who have received their last dT(Pa) vaccine at least 5 years ago, and who have the Visit 2 on 'Day 2'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 2 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Placebo (Saline)
- Placebo, Female, >/= 5 years, D3 visit (Placebo Comparator): 5 female subjects who have received their last dT(Pa) vaccine at least 5 years ago, and who have the Visit 2 on 'Day 3'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Placebo (Saline)
- Boostrix, Male, <5 years, D2 visit (Active Comparator): 25 male subjects who have received their last dT(Pa) vaccine between 5 years and 6 months ago, and who have the Visit 2 on 'Day 2'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 2 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Boostrix
- Boostrix, Male, <5 years, D3 visit (Active Comparator): 25 male subjects who have received their last dT(Pa) vaccine between 5 years and 6 months ago, and who have the Visit 2 on 'Day 3'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Boostrix
- Boostrix, Female, <5 years, D2 visit (Active Comparator): 25 female subjects who have received their last dT(Pa) vaccine between 5 years and 6 months ago, and who have the Visit 2 on 'Day 2'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 2 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Boostrix
- Boostrix, Female, <5 years, D3 visit (Active Comparator): 25 female subjects who have received their last dT(Pa) vaccine between 5 years and 6 months ago, and who have the Visit 2 on 'Day 3'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Boostrix
- Placebo, Male, <5 years, D2 visit (Placebo Comparator): 5 male subjects who have received their last dT(Pa) vaccine between 5 years and 6 months ago, and who have the Visit 2 on 'Day 2'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 2 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Placebo (Saline)
- Placebo, Male, <5 years, D3 visit (Placebo Comparator): 5 male subjects who have received their last dT(Pa) vaccine between 5 years and 6 months ago, and who have the Visit 2 on 'Day 3'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Placebo (Saline)
- Placebo, Female, <5 years, D2 visit (Placebo Comparator): 5 female subjects who have received their last dT(Pa) vaccine between 5 years and 6 months ago, and who have the Visit 2 on 'Day 2'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 2 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Placebo (Saline)
- Placebo, Female, <5 years, D3 visit (Placebo Comparator): 5 female subjects who have received their last dT(Pa) vaccine between 5 years and 6 months ago, and who have the Visit 2 on 'Day 3'.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 28 (blood sampling)
  Interventions: Biological: Placebo (Saline)

INTERVENTIONS:
Biological: Boostrix — Randomised assignment
  Arms: Boostrix, Female, <5 years, D2 visit; Boostrix, Female, <5 years, D3 visit; Boostrix, Female, >/= 5 years, D2 visit; Boostrix, Female, >/= 5 years, D3 visit; Boostrix, Male, <5 years, D2 visit; Boostrix, Male, <5 years, D3 visit; Boostrix, Male, >/= 5 years, D2 visit; Boostrix, Male, >/= 5 years, D3 visit
Biological: Placebo (Saline) — Randomised assignment
  Arms: Placebo, Female, <5 years, D2 visit; Placebo, Female, <5 years, D3 visit; Placebo, Female, >/= 5 years, D2 visit; Placebo, Female, >/= 5 years, D3 visit; Placebo, Male, <5 years, D2 visit; Placebo, Male, <5 years, D3 visit; Placebo, Male, >/= 5 years, D2 visit; Placebo, Male, >/= 5 years, D3 visit

SUMMARY:
The purpose of this protocol is to generate a set of data that will be analysed by integrated systems biology approach, for validation in subsequent clinical trials or in animal models.

240 healthy participants (18-45y) will be enrolled, 200 will be administered a dose of Boostrix on Day 0, 20 will receive a placebo on Day 0.

DETAILED DESCRIPTION:
This study is part of the BIOVACSAFE project, a 5-year project funded by the Innovative Medicine Initiative, which will undertake a series of correlated clinical studies that will apply and develop technologies to generate clinical data on inflammation with licensed vaccines as benchmarks, and identify biomarkers to predict acceptable reactogenicity, for correlation with standardized clinical readouts and inflammatory markers assessed in natural infections.

The purpose of this protocol is to generate data to undergo integrated systems biology analysis to validate biomarkers identified in the exploratory studies conducted previously or to identify new biomarkers of responses to immunisation

The data set will include data characterising:

1. Physiological responses at various time points after immunisation by measuring:

   * Local and systemic vaccine-related clinical events.
   * Haematology (blood counts and ESR) and biochemistry parameters.
2. Innate and adaptive immune responses including:

   * Innate immune activation detected by global gene expression in whole blood
   * Adaptive humoral immunity determined by the quantification antibodies directed against Tetanus toxoid (TT), Diphteria toxoid (DT), Pertussis toxin (PT), Fimbrial haemagglutinin (FHA) and Pertactin (PTN).
   * Adaptive immune activation detected by gene pathway activation in whole blood
   * Metabolic responses as detected by metabolic gene expression and pathway activation in whole blood
   * Innate and adaptive immune activation detected by measuring the concentration of selected soluble mediators in serum including: chemokines and cytokines and acute phase proteins
   * As an exploratory endpoint, the adaptive cellular immune response will be evaluated via counting vaccine antigen-specific Cluster of Differentiation 4 (CD4)+ T cells expressing activation markers and/or cytokines following in vitro stimulation and analysis by flow cytometry (and or CyTOF).
3. Genetic testing of subjects when deemed necessary (genetic testing analysis may be SNP (single nucleotide polymorphism) analysis or full genome analysis).
4. Correlations in changes in innate immune activation and metabolism with adverse events, haematology and biochemistry panels, genotype and physiological assessments

The investigators will biobank all samples for the duration of the BIOVACSAFE programme so that they can selectively analyse different samples and different time points depending on the results generated, principally from the gene expression analysis of whole blood.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18-45 years (inclusive).
2. Male: Female ratio - 1:1.
3. Half of the subjects (n=120) will have received a previous Dt(pa) dose less than 5 years before, the other half (n=120) will have received a previous Dt(pa) dose 5 or more years before participating at this study.
4. The subject is, in the opinion of the investigator healthy based on medical history and clinical exam, with no active disease process that could interfere with the study endpoints.
5. Has a body Mass Index ≥18.0 and ≤30.0
6. Is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
7. The subject has signed the ICF.
8. The subject is available for follow-up for the duration of the study.
9. The subject agrees to abstain from donating blood during their participation in the study, or longer if necessary.
10. If the subject is a heterosexually active female, she is willing to use an effective method of contraception with partner (oral contraceptive pill; intrauterine device; injectable or implanted contraceptive; condoms incorporating spermicide if using these; physiological or anatomical sterility) from 30 days prior to, and 3 months after, vaccination. Willing to undergo urine pregnancy tests prior to vaccination at screening.
11. The subject has venous access sufficient to allow blood sampling as per the protocol.

    Exclusion Criteria:
12. Pregnant or lactating at any point during the study from screening to final follow up.
13. Hypersensitivity to any component of the vaccine or subjects having shown signs of hypersensitivity after previous administration of diphtheria, tetanus, or pertussis vaccines.
14. Presence of primary or acquired immunodeficiency states with a total lymphocyte count less than 1,200 per mm3 or presenting other evidence of lack of cellular immune competence e.g. leukaemias, lymphomas, blood dyscrasias, or patients receiving immunosuppressive therapy (including regular use of oral or parenteral corticosteroids).
15. Use of any immune suppressing or immunomodulating drugs within 6 months of Visit 1.
16. Regular and prolonged use of non-steroidal anti-inflammatory drugs (oral or parenteral route) within 6 months of Visit 1 considered by the study physician as likely to interfere with immune responses.
17. Current intake of excessive amounts of alcohol and/or caffeine (as evaluated by the investigator) and not willing to adapt this use during the study period.
18. Currently performing extreme physical activities (as evaluated by the investigator) and not willing to adapt this use during the study period.
19. Receipt of a vaccine within 30 days prior to visit 1, or requirement to receive a vaccine within the 28 days following study vaccination, vaccination with a tetanus, diphtheria, pertussis combined vaccine within the last 6 months before the first study visit.
20. Presence of an acute severe febrile illness at time of immunisation.
21. History of alcohol, narcotic, benzodiazepine, rilatine, or other substance abuse or dependence within the 12 months preceding Visit 1.
22. Currently participating in another clinical study with an investigational or non-investigational drug or device, or has participated in a clinical trial within the 3 months preceding Visit 1.
23. Any condition that, in the investigator's opinion, compromises the subject's ability to meet protocol requirements or to complete the study.
24. Receipt of blood products or immunoglobulins, or blood donation within 3 months prior to visit 1.
25. Unable to read and speak Dutch or English to a fluency level adequate for the full comprehension of procedures required in participation and consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Frequency of local vaccine-related clinical events | At all timepoints from vaccination up to 28 days after vaccination
  Participants will report these events on a diary, measuring local events or scoring them from 0 (absent) to 3 (severe)
Frequency of systemic vaccine-related clinical events. | At all timepoints from vaccination up to 28 days after vaccination
  Participants will report these events on a diary, scoring them from 0 (absent) to 3 (severe)
Physiological assessments: Change from pre-immunisation baseline values in body temperature. | Up to 7 days after vaccination
Change from pre-immunisation baseline values in 'Erythrocyte Sedimentation Rate' (ESR) | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in creatinin | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in C Reactive Protein (CRP) | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in aspartate transaminase (AST)/ alanine transaminase (ALT) | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in albumin | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in estimated glomerular filtration rate (eGFR) | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in gamma glutamyl transpeptidase (GGT) | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in total protein | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in prothrombin/fibrinogen | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in global gene expression measured on whole blood samples. | At selected timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in metabolic gene expression measured on whole blood samples. | At selected timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in serum levels of antibodies to vaccine antigens (anti-T, anti-D, anti-PT, anti-FHA and anti-PRN) in serum samples. | At selected timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation values of adaptive cellular immune response via enumeration of TT-, DT-, PT-, FHA- and PTN-specific CD3/CD4+ or CD3/CD8+ T cells expressing activation markers/cytokines following IV stimulation and analysis by flow cytometry. | At 7 days after vaccination
Change from pre-immunisation baseline values in concentration of selected cytokines and acute phase proteins in serum samples | At selected timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in pathway activation measured on whole blood samples. | At selected timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in haemoglobin | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in red blood cell count | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in haematocrit | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in white blood cell count | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in platelet count | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in white blood cells | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in 'mean corpuscular volume' | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in 'mean corpuscular heamoglobin' | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in 'mean corpuscular heamoglobin concentration' | At all timepoints from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in Cell Mediated Immunity status in response to in vitro antigen stimulation | At all timepoints from vaccination up to 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Geert Leroux-Roels, Prof., MD, Principal Investigator — Center for Vaccinology
Locations (1):
- Center for Vaccinology, Ghent, East-Flanders, Belgium